CLINICAL TRIAL: NCT00952341
Title: A Phase III, Randomized, Multi-center, Double-Blind, Placebo-Controlled, Parallel-Group Clinical Trial to Study the Safety, Tolerability and Efficacy of MK0869/Aprepitant for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) Associated With High-Dose Cisplatin
Brief Title: Aprepitant/MK0869 for Prevention of Chemotherapy Induced Nausea and Vomiting Associated With Cisplatin (0869-169)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0869-169; 2009_626
Record Dates: First submitted 2009-07-31; First posted 2009-08-06 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Chemotherapy-induced Nausea and Vomiting (CINV)
Keywords: CINV
MeSH Terms: conditions — Vomiting | interventions — Aprepitant; Dexamethasone; Granisetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant (MK-0869) (Experimental)
  Interventions: Drug: aprepitant; Drug: granisetron; Drug: dexamethasone
- Standard Therapy (Placebo Comparator)
  Interventions: Drug: Comparator: Placebo to aprepitant; Drug: dexamethasone; Drug: granisetron

INTERVENTIONS:
Drug: aprepitant — Day 1: Oral aprepitant 125 mg prior to administration of cisplatin; Days 2 and 3: Oral aprepitant 80 mg
  Arms: Aprepitant (MK-0869)
Drug: Comparator: Placebo to aprepitant — Day 1: Placebo to oral aprepitant 125 mg prior to administration of cisplatin; Days 2 and 3: Placebo to oral aprepitant 80 mg
  Arms: Standard Therapy
Drug: dexamethasone — Day 1: Oral dexamethasone 10.5 mg prior to administration of cisplatin; Days 2, 3, and 4: Oral dexamethasone 7.5 mg
  Arms: Standard Therapy
Drug: granisetron — Day 1: IV granisetron 3 mg prior to administration of cisplatin
Drug: dexamethasone — Day 1: oral dexamethasone 6 mg prior to the administration of cisplatin; Days 2 and 3: oral dexamethasone 3.75 mg
  Arms: Aprepitant (MK-0869)

SUMMARY:
This study will demonstrate and confirm the efficacy and safety of MK0869 for the treatment of chemotherapy-induced nausea and vomiting in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

Cycle 1:

* Patient is scheduled to receive his/her first course of cisplatin chemotherapy at a dose of at least 70 mg/m^2 administered a maximum of 3 hours
* Patient has a predicted life expectancy of at least 3 months
* Patient is not pregnant

Cycle 2 (optional):

* Participation in the study during the next cycle of chemotherapy is considered

appropriate by the investigator and will not pose unwarranted risk to the patient.

* Satisfactory completion of the preceding cycle of chemotherapy and related

study procedures.

* Patient will continue to receive the same chemotherapy regimen as in Cycle 1. The cisplatin dose may be reduced in subsequent cycle, as long as the new

dose is still no less than 70 mg/m^2.

Exclusion Criteria:

Cycles 1 & 2:

* Patient will receive stem cell therapy in conjunction with cisplatin
* Patient has an active infection or any uncontrolled disease (e.g. diabetes)
* Patient will receive multiple-day chemotherapy with cisplatin
* Patient will receive chemotherapy of moderate or high emetogenicity on the 6 days prior to cisplatin infusion or the 6 days following the cisplatin infusion
* Patient has vomited within 24 hours prior to cisplatin infusion
* Patient received or will receive radiation therapy to the abdomen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2009-08-25 (Actual); Primary Completion 2010-04-04 (Actual); Study Completion 2010-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hu Z, Cheng Y, Zhang H, Zhou C, Han B, Zhang Y, Huang C, Chang J, Song X, Liang J, Liang H, Bai C, Yu S, Chen J, Wang J, Pan H, Chitkara DK, Hille DA, Zhang L. Aprepitant triple therapy for the prevention of chemotherapy-induced nausea and vomiting following high-dose cisplatin in Chinese patients: a randomized, double-blind, placebo-controlled phase III trial. Support Care Cancer. 2014 Apr;22(4):979-87. doi: 10.1007/s00520-013-2043-9. Epub 2013 Nov 26. PMID 24276953

RESULTS

PARTICIPANT FLOW:
Groups:
- Aprepitant (MK-0869): Day 1: Oral aprepitant 125 mg prior to administration of cisplatin; Days 2 and 3: Oral aprepitant 80 mg
  Day 1: Intravenous (IV) granisetron 3 mg prior to administration of cisplatin
  Day 1: oral dexamethasone 6 mg prior to the administration of cisplatin; Days 2 and 3: oral dexamethasone 3.75 mg
- Placebo: Day 1: Placebo to oral aprepitant 125 mg prior to administration of cisplatin; Days 2 and 3: Placebo to oral aprepitant 80 mg
  Day 1: Oral dexamethasone 10.5 mg prior to administration of cisplatin; Days 2, 3, and 4: Oral dexamethasone 7.5 mg
  Day 1: IV granisetron 3 mg prior to administration of cisplatin
Period: Cycle 1
Arm/Group | Aprepitant (MK-0869) | Placebo
Started | 209 | 212
Completed | 189 | 199
Not Completed | 20 | 13
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Protocol Violation | 2 | 1
Not completed — Lost to Follow-up | 11 | 2
Not completed — Physician Decision | 0 | 1
Period: Cycle 2
Arm/Group | Aprepitant (MK-0869) | Placebo
Started | 110 | 130
Completed | 101 | 118
Not Completed | 9 | 12
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 6 | 9
Not completed — Physician Decision | 1 | 1
Not completed — Progressive Disease | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant (MK-0869) | Placebo | Total
Number analyzed (Participants) | 209 | 212 | 421
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (10.1) | 53.6 (10.6) | 53.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 73 | 144
  Male | 138 | 139 | 277
Region of Enrollment [Number; unit: participants]
  China | 209 | 212 | 421

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Complete Response 120 Hours Following Initiation of High-dose Cisplatin Chemotherapy in the Overall Phase of Cycle 1
Description: Overall phase was defined as 0 to 120 hours following initiation of chemotherapy.
  Complete response was defined as no vomiting with no rescue therapy.
Time Frame: 0 to 120 hours
Population: Full Analysis Set (FAS), defined as those who received chemotherapy, received a dose of study drug and had at least one post-treatment assessment. Any participant who did not have a response recorded for the assessment was excluded from the analysis.
Measure: Number; unit: Proportion of participants
Arm/Group | Aprepitant (MK-0869) | Placebo
Number analyzed (Participants) | 204 | 207
Proportion of participants | 0.696 | 0.570
Statistical Analysis 1: Comparison: Aprepitant (MK-0869) vs Placebo; Adjusted by gender and concomitant chemotherapy. The apriori significance level was set at 0.05. There was no adjustment for multiplicity; Test type: Superiority or Other; p = 0.007, Regression, Logistic

2. Secondary Outcome: Proportion of Participants With Complete Response in the Acute Phase of Cycle 1
Description: Acute phase was defined as 0 to 24 hours following initiation of chemotherapy.
  Complete response was defined as no vomiting with no rescue therapy.
Time Frame: 0 to 24 hours
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Aprepitant (MK-0869) | Placebo
Number analyzed (Participants) | 204 | 208
Proportion of participants | 0.794 | 0.793
Statistical Analysis 1: Comparison: Aprepitant (MK-0869) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.942, Regression, Logistic

3. Secondary Outcome: Proportion of Participants With Complete Response in the Delayed Phase of Cycle 1
Description: Delayed phase was defined as 25 to 120 hours following initiation of chemotherapy.
  Complete response was defined as no vomiting with no rescue therapy.
Time Frame: 25 to 120 hours
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Aprepitant (MK-0869) | Placebo
Number analyzed (Participants) | 204 | 207
Proportion of participants | 0.740 | 0.594
Statistical Analysis 1: Comparison: Aprepitant (MK-0869) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, Regression, Logistic

4. Secondary Outcome: Proportion of Participants With No Vomiting in the Overall Phase of Cycle 1
Description: Overall Phase was defined as 0 to 120 hours following initiation of chemotherapy.
  No vomiting was defined as no vomiting or retching or dry heaves (included participants who received rescue therapy).
Time Frame: 0 to 120 hours
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Aprepitant (MK-0869) | Placebo
Number analyzed (Participants) | 204 | 207
Proportion of participants | 0.706 | 0.570
Statistical Analysis 1: Comparison: Aprepitant (MK-0869) vs Placebo; Adjusted by gender and concomitant chemotherapy; Test type: Superiority or Other; p = 0.003, Regression, Logistic

5. Secondary Outcome: Proportion of Participants With No Vomiting in the Acute Phase of Cycle 1
Description: Acute Phase was defined as 0 to 24 hours following initiation of chemotherapy.
Time Frame: 0 to 24 hours
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Aprepitant (MK-0869) | Placebo
Number analyzed (Participants) | 204 | 208
Proportion of participants | 0.804 | 0.798
Statistical Analysis 1: Comparison: Aprepitant (MK-0869) vs Placebo; Adjusted by gender and concomitant chemotherapy; Test type: Superiority or Other; p = 0.882, Regression, Logistic

6. Secondary Outcome: Proportion of Participants With No Vomiting in the Delayed Phase of Cycle 1
Description: Delayed Phase was defined as 25 to 120 hours following initiation of chemotherapy
Time Frame: 25 to 120 hours
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Aprepitant (MK-0869) | Placebo
Number analyzed (Participants) | 204 | 207
Proportion of participants | 0.740 | 0.594
Statistical Analysis 1: Comparison: Aprepitant (MK-0869) vs Placebo; Adjusted by gender and concomitant chemotherapy; Test type: Superiority or Other; p = 0.001, Regression, Logistic

7. Secondary Outcome: Proportion of Participants With No Impact on Daily Life in Cycle 1
Description: The Functional Living Index-Emesis is a self-administered, validated emesis & nausea-specific questionnaire. Participants completed the questionnaire 5 days post chemotherapy. It had 9 questions each on nausea and vomiting. "No impact of chemotherapy-induced nausea & vomiting (CINV) on daily life" was defined as an average item score of >6 on the 7-point scale (i.e., >108 total score). The scale was in the opposite direction for questions 3, 6, 11, 15 & 18. For each question: score ranged from 1 (worst) to 7 (best, i.e., no CINV). Total score range was 7 (worst) to 126 (best).
Time Frame: 0 to 120 hours
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Aprepitant (MK-0869) | Placebo
Number analyzed (Participants) | 200 | 202
Proportion of participants | 0.705 | 0.683

8. Secondary Outcome: Time to First Vomiting Episode in Cycle 1
Description: Time from administration of chemotherapy to first vomiting episode.
Time Frame: 0 to 120 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Aprepitant (MK-0869) | Placebo
Number analyzed (Participants) | 204 | 207
Hours | 77.0 (2.5) | 76.0 (2.8)

ADVERSE EVENTS:
Description: The All Patients as Treated (APaT) population were used for the analysis of
  safety data in this study. The APaT population consisted of all randomized patients who received at least one dose of study medication.
Groups:
- Aprepitant (MK-0869), Cycle 1 & Cycle 2: Day 1: Oral aprepitant 125 mg prior to administration of cisplatin; Days 2 and 3: Oral aprepitant 80 mg
  Day 1: IV granisetron 3 mg prior to administration of cisplatin
  Day 1: oral dexamethasone 6 mg prior to the administration of cisplatin; Days 2 and 3: oral dexamethasone 3.75 mg
- Placebo, Cycle 1 & Cycle 2: Day 1: Placebo to oral aprepitant 125 mg prior to administration of cisplatin; Days 2 and 3: Placebo to oral aprepitant 80 mg
  Day 1: Oral dexamethasone 10.5 mg prior to administration of cisplatin; Days 2, 3, and 4: Oral dexamethasone 7.5 mg
  Day 1: IV granisetron 3 mg prior to administration of cisplatin
Arm/Group | Aprepitant (MK-0869), Cycle 1 & Cycle 2 | Placebo, Cycle 1 & Cycle 2
Serious Adverse Events (participants affected / at risk) | 5/205 | 2/210
Other Adverse Events (participants affected / at risk) | 123/205 | 124/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant (MK-0869), Cycle 1 & Cycle 2 (N=205) | Placebo, Cycle 1 & Cycle 2 (N=210)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant (MK-0869), Cycle 1 & Cycle 2 (N=205) | Placebo, Cycle 1 & Cycle 2 (N=210)
Constipation (Gastrointestinal disorders) | 38 (41) | 31 (37)
Diarrhoea (Gastrointestinal disorders) | 13 (13) | 8 (8)
Nausea (Gastrointestinal disorders) | 12 (12) | 21 (22)
Vomiting (Gastrointestinal disorders) | 7 (7) | 29 (31)
Fatigue (General disorders) | 13 (14) | 4 (4)
Pyrexia (General disorders) | 11 (13) | 5 (5)
Alanine aminotransferase increased (Investigations) | 20 (22) | 21 (27)
Aspartate aminotransferase increased (Investigations) | 7 (8) | 11 (12)
Haemoglobin decreased (Investigations) | 15 (17) | 11 (16)
Neutrophil count decreased (Investigations) | 33 (42) | 39 (48)
White blood cell count decreased (Investigations) | 50 (65) | 49 (61)
Decreased appetite (Metabolism and nutrition disorders) | 30 (33) | 29 (32)
Insomnia (Psychiatric disorders) | 5 (5) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.